CLINICAL TRIAL: NCT02343627
Title: A Randomized, Double-Blind, Placebo-Controlled, Pilot Study to Assess the Safety and Efficacy of NVXT Solution in Patients With Mild-to-Moderate Fungal Infection of the Toe Nail
Brief Title: Safety and Efficacy of NVXT Solution in Mild-to-Moderate Fungal Infection of the Toe Nail
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sun Pharmaceutical Industries, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NVXT 1405
Record Dates: First submitted 2014-12-27; First posted 2015-01-22 (Estimated); Results first posted 2018-08-22 (Actual); Last update posted 2018-09-19 (Actual); Status verified 2018-08

CONDITIONS: Onychomycosis
MeSH Terms: conditions — Onychomycosis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- NVXT Solution (Experimental): NVXT Solution once daily for 60 days
  Interventions: Drug: NVXT Solution
- Vehicle of test product (Placebo Comparator): Vehicle of test product, once daily for 60 days
  Interventions: Drug: Vehicle of test product

INTERVENTIONS:
Drug: NVXT Solution — NVXT Solution, applied to infected toe nails and 0.5 mm of adjacent skin once daily for 60 days.
  Other Names: NVXT
  Arms: NVXT Solution
Drug: Vehicle of test product — Vehicle of test product applied to infected toe nails and 0.5 mm of adjacent skin once daily for 60 days.
  Other Names: Placebo
  Arms: Vehicle of test product

SUMMARY:
This study will examine the safety, tolerability and efficacy of NVXT in a new formulation in patients with mild-to-moderate fungal infection of the toe nail.

DETAILED DESCRIPTION:
This Phase IIa pilot multiple-dose study will examine the safety, tolerability and efficacy of NVXT in a new formulation in patients with mild-to-moderate fungal infection of the toe nail.

ELIGIBILITY:
Inclusion Criteria:

* Clinically diagnosed onychomycosis
* Presence of dermatophyte fungal infection with no current topical or systemic antifungal therapy
* Clinical diagnosis of mild-to-moderate fungal infection of at least one toe involving 10-50% of the nail area, without involvement of one of the lunular proximal regions
* Positive potassium hydroxide mount preparation
* Positive fungal culture for a dermatophyte

Exclusion Criteria:

* Nail or anatomical abnormalities of the toe that may interfere with evaluations or dosing compliance

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2014-12; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Taro Pharmaceuticals USA, Study Director — Taro Pharmaceuticals USA Inc.

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | NVXT Solution | Vehicle of Test Product
Started | 35 | 12
Completed | 23 | 11
Not Completed | 12 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | NVXT Solution | Vehicle of Test Product | Total
Number analyzed (Participants) | 35 | 12 | 47
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 35 | 12 | 47
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 1 | 6
  Male | 30 | 11 | 41
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 9 | 5 | 14
  White | 21 | 5 | 26
  More than one race | 5 | 2 | 7
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Negative Fungal Culture
Description: To assess number of participants with negative fungal culture after repeated once-daily topical applications for 28 days
Time Frame: 28 days
Population: Subjects with fungal culture collected at the study day 28 visit. The subjects may not complete all study visits.
Measure: Count of Participants; unit: Participants
Arm/Group | NVXT Solution | Vehicle of Test Product
Number analyzed (Participants) | 33 | 12
Participants | 14 | 2

ADVERSE EVENTS:
Arm/Group | NVXT Solution | Vehicle of Test Product
Serious Adverse Events (participants affected / at risk) | 0/35 | 0/12
Other Adverse Events (participants affected / at risk) | 7/35 | 3/12
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | NVXT Solution (N=35) | Vehicle of Test Product (N=12)
Hypertension (Vascular disorders) | 0 (0) | 1 (1)
Abdominal Pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Common Cold (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Pharangitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Sinusitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Muscle Spasm (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Exacerbation of Tinea Pedis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No